CLINICAL TRIAL: NCT06954350
Title: Investigation of Pain, Sleep Quality, Eating Habits and Physical Activity Level in Patients With Bipolar Disorder in Euthymic Period
Brief Title: Pain, Sleep Quality, Eating Habits and Physical Activity Level in Patients With Bipolar Disorder
Status: Enrolling by invitation | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Vedat KURT, Assos. Prof., Kutahya Health Sciences University
Other Study IDs: 2024/14-10
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Bipolar Disorder (BD)
Keywords: Bipolar Disorder; Pain; Sleep Quality
MeSH Terms: conditions — Bipolar Disorder; Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bipolar disorder (BD) is a complex condition characterized by recurrence of mania, hypomania, and depression. It is characterized by changes in daily life activities, sleep status, focus problems, and cognitive fluctuations. The mortality rate due to suicide and cardiovascular diseases increases in individuals with BD. The DSM-5TR defines BD as Bipolar I Disorder (BD-1) with one or more manic episodes, Bipolar II Disorder (BD-II) with at least one severe depressive episode accompanied by at least one hypomanic episode, Cyclothymia disorder, substance-induced bipolar disorder, bipolar or related disorder related to another medical condition, other defined bipolar and related disorder, and undefined bipolar and related disorder. The lifetime prevalence of BD varies between 0.6% and 1.0% for Type I and 0.4% and 1.1% for Type II. Symptoms usually start between 14-21 years of age. Depressive episodes and lifelong single marital status are more common in females, while substance abuse is more common in males.

Depression attacks are longer than manias, but the duration of attacks does not differ between types. The mean duration of depressive and manic periods is 5.2 months and 3.5 months, respectively. Pain is observed in 28.9% of patients with a diagnosis of GI, which decreases the quality of life and is a significant concern in psychological disorders.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is assumed to be a multifactorial entity including psychosocial and genetic factors whose neurobiology is still unclear. BD is characterised by recurrence of mania, hypomania and depression. In the fluctuations seen in these transitions, individuals may experience changes in daily life activities and sleep status, focussing problems and cognitive fluctuations. The mortality rate due to suicide and cardiovascular diseases increases in individuals with BD. DSM-5TR defines BD as Bipolar I Disorder (BD-1) in the presence of one or more manic episodes, Bipolar II Disorder (BD-II) in the presence of at least one severe depressive episode accompanied by at least one hypomanic episode, Cyclothymia disorder which does not meet the criteria for BD I-II but has a course closer to normal including prolonged hypomanic and depressive episodes, It is classified as substance-induced bipolar disorder which occurs in case of intoxication or withdrawal as a result of the use of drugs or medications, bipolar or related disorder related to another medical condition, other defined bipolar and related disorder including mild and atypical symptoms, and undefined bipolar and related disorder in which symptoms are predominant but diagnostic criteria are not sufficiently present.

The lifetime prevalence of BD is estimated to vary between 0.6% and 1.0% for Type I and between 0.4% and 1.1% for Type II. Symptoms of most of the cases start between 14-21 years of age. Although there are no major differences between genders, depressive episodes and lifelong single marital status are more common in female individuals and substance abuse is more common in male individuals.

In a study examining the duration of attacks, it was reported that depression attacks were much longer than manias, but the duration of attacks did not differ between types and the mean duration of depressive and manic periods were 5.2 months and 3.5 months, respectively. In the manic period, the level of consciousness of the patients is generally clear and attention is increased. However, clouding of consciousness may occur due to reasons such as being physically more active than normal and disrupting or reducing eating patterns. Sudden sleep disturbances such as difficulty falling asleep and waking up at unusual hours may be a sign of mania. Excessive physical activity may cause exhaustion and weight loss with the emergence of nutritional problems. Although consciousness is intact during depression, blurred consciousness may occur in exhausted and numbness depressions. Increased desire for sleep, decreased appetite, exhaustion and decreased sexual desire may be observed.

Pain is observed in 28.9% of patients with a diagnosis of GI. The prevalence of pain in patients, especially chronic pain and migraine, decreases the quality of life and studies in this patient group are limited. Acute pain, on the other hand, has been shown in one study to be 83% of those who felt pain momentarily. Since chronic pain triggers recurrent thoughts of death, pain management should be a part of treatment in psychological disorders.

In the literature, quality of life, sleep disorder, eating disorder, physical activity, suicidal ideation and pain (localisation and intensity) of patients diagnosed with bipolar disorder have been examined separately, but there are few studies on pain in bipolar disorder. In our country, it is observed that there have not been many studies on pain assessment in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 65.
* Being diagnosed with bipolar disorder by a psychiatrist according to DSM-5 criteria and not having symptoms of depression and mania at a level that prevents participation in the study.
* Volunteering to participate in the study.

Exclusion Criteria:

* Not being able to read and write Turkish.
* Having mental retardation.
* Having suffered a severe head trauma in the last 1 year.
* Having a disease that affects cognitive functions such as dementia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Being diagnosed with bipolar disorder
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Pain Intensty | at enrollment
  The McGill Pain Questionnaire consists primarily of 3 major classes of word descriptors--sensory, affective and evaluative--that are used by patients to specify subjective pain experience. It also contains an intensity scale and other items to determine the properties of pain experience. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
Pain quality and type | At enrollment
  To assess pain quality and type, participants were asked to choose as many of the words as possible from a list containing 29 adjectives of pain sensation descriptors taken from the McGill Pain Questionnaire (MPQ). Sensations of shooting, stabbing, electric shock-like, nagging, numbness, tingling, and burning were considered as neuropathic pain descriptors, whereas non-neuropathic pain was described as a sharp, aching, or throbbing sensation. Superficial pain descriptors included numbness, tingling, burning, shooting, sharp, pressure, piercing, stinging, hot, smarting, radiating, and cutting, while deep pain descriptors included cramping, tenderness, aching, pulling, pounding, gnawing, soreness, boring, stabbing, troublesome, annoying, dull, nagging, and throbbing.
Pain distribution | At enrollment
  Pain distribution was measured using the Margolis drawing rating system, which has 45 anatomical areas, each with a corresponding percentage value of body surface, in order to compute a total weighted score, indicating body pain distribution.

SECONDARY OUTCOMES:
Pittsburgh sleep quality index | At enrollment
  The questionnaire has a blend of Likert-type and open-ended questions, which are subsequently transformed into scaled scores according to the provided standards.
  Participants are requested to specify the frequency of their sleep difficulties encountered in the preceding month and to evaluate their overall sleep quality.Values for each item vary from 0 to 3, with elevated values signifying more severe sleep disruptions.Developers proposed a threshold score of 5 for the global scale, since it accurately identified 88.5% of the patient cohort in their validation research.

CONTACTS AND LOCATIONS:
Locations (1):
- Helath Sciences Faculty, Kütahya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided